CLINICAL TRIAL: NCT03962361
Title: New Biomarkers of Neurological Outcome in Patients With Sudden Cardiac Death: Role of Circulating Microparticles
Brief Title: New Biomarkers of Neurological Outcome After a Sudden Cardiac Death
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBPS-BIO-2015-56
Record Dates: First submitted 2016-06-13; First posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Cardiac Sudden Death; Hypoxia Brain; Cell Membrane Microparticles; Biomarkers
Keywords: Cardiac Sudden Death; Hypoxia Brain; Biomarkers; Cell-Derived Microparticles
MeSH Terms: conditions — Death, Sudden, Cardiac; Hypoxia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood samples from patients enrolled in the study will be collected at admission, at 24 and at 72 hours. Blood collection will be obtained from arterial access whenever possible (otherwise preferably central or peripheral venous lines will be used without using tourniquet) and stored in tubes sodium citrate 3.8 %. Immediately after blood collection, the proteolipid protein fraction will be obtained by centrifugation fraction. To do this , samples will be centrifuged twice to exclude any cell rest. The aliquots obtained will be frozen first with liquid nitrogen and then stored at -80°C in the Biobank IIB Sant Pau until further analysis.

GROUPS / COHORTS (1):
- Sudden cardiac death of ischemic cause: Patients admitted to the Coronary Care Unit for sudden cardiac death of ischemic cause and remain comatose (GCS < 8 points).
  Interventions: Other: Concentration of circulating microparticles.

INTERVENTIONS:
Other: Concentration of circulating microparticles. — The microparticles contained in the blood sample will be isolated by ultracentrifugation and quantified by flow cytometry. The microparticles concentration will be determined by the number of microparticles per uL of plasma, based on the volume of the sample, the flow rate of the cytometer and the number of fluorescent events.

SUMMARY:
The aim of the project is to establish the value of circulating microparticles as a new biomarker for neurological prognosis of patients recovered from sudden cardiac death who remain comatose.

DETAILED DESCRIPTION:
This is a pilot study. Analytical, observational, longitudinal, retrospective and prospective, non-randomized. Patients recovered from sudden cardiac death of ischemic cause and remain comatose will be included in the protocol if they fit the pre-specified inclusion criteria. Biological samples will be collected (at admission, at 24 and 72 hours) and stored in the Biobank of Hospital de la Santa Creu i Sant Pau for further analysis. In addition demographic, clinical and analytical variables will be collected. At the end of the recruitment period, we will analyse the concentrations of circulating microparticles according to ICCC-IIBSantPau methodology in the samples obtained. The primary outcome variable will be the neurological status at Coronary Care Unit discharge and at 6 months. The objective of the study will evaluate the relationship between the neurological status and the blood concentrations of circulating microparticles.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old.
* Patients recovered from a sudden cardiac death (in-hospital and out-of-hospital) with return of spontaneous circulation (ROSC) (defined as systolic blood pressure > 60 mmHg or palpable pulse for > 5 minutes) who remain unconsciousness (defined as a score on the Glasgow Coma Scale <8 ) for > 5-10 minutes after ROSC.
* Treated with hypothermia as recommended by the European guidelines for resuscitation ( 2010)..

Exclusion Criteria:

* Non-cardiac sudden death.
* Active oncologic pathology .
* Traumatic or spontaneous intra-cranial haemorrhage.
* Inability to obtain required blood samples or refusal of the informed consent necessary for it.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will include patients who have suffered a sudden cardiac death of ischemic cause admitted to the Coronary Care Unit of the Hospital de la Santa Creu i Sant Pau in Barcelona from the date of commencement of the study. The sample will be retrospectively completed with patients of the same features admitted to the unit since January 2012 and who have biological samples stored in the Biobank of Hospital de la Santa Creu i Sant Pau.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2016-02; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in Glasgow-Pittsburgh Cerebral Performance Categories Scale for neurological outcome. | Change from Glasgow-Pittsburgh Cerebral Performance Categories Scale at 6 months
  1. Good cerebral performance: conscious, alert, able to work, might have mild neurologic or psychologic deficit.
  2. Moderate cerebral disability: conscious, sufficient cerebral function for independent activities of daily life. Able to work in sheltered environment.
  3. Severe cerebral disability: conscious, dependent on others for daily support because of impaired brain function. Ranges from ambulatory state to severe dementia or paralysis.
  4. Coma or vegetative state: any degree of coma without the presence of all brain death criteria. Unawareness, even if appears awake (vegetative state) without interaction with environment; may have spontaneous eye opening and sleep/awake cycles. Cerebral unresponsiveness.
  5. Brain death: apnea, areflexia, EEG silence, etc.

SECONDARY OUTCOMES:
Cardiovascular mortality | 6 months
  Cardiovascular mortality

CONTACTS AND LOCATIONS:
Overall Officials: Laia C Belarte, Doctor, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain